

## Pilot Study for Investigating the Effect of the Bruder Eye Hydrating Compress on Contact Lens Discomfort in Contact Lens Wearers

## **Statistical Plan**

PRINCIPAL INVESTIGATOR:

JASON J. NICHOLS, OD MPH PhD

**CO-INVESTIGATOR:** 

ANNA F. ABLAMOWICZ, OD

UNIVERSITY OF ALABAMA AT BIRMINGHAM

**SCHOOL OF OPTOMETRY** 

1716 UNIVERSITY BLVD

**BIRMINGHAM, AL 35294-0010** 

## Statistical Analyses

Descriptive statistics will be performed and differences in groups at baseline analyzed using the Kruskal-Wallis test and the Chi-square test for categorical variables. Statistical testing of the primary endpoint will be performed using a generalized linear model with treatment and baseline as main effects while controlling for difference in comfortable wear time at baseline and daily hours of contact lens wear time. A one-way analysis of variance (ANOVA) will be used to compare the mean hours of comfortable contact lens wear time at 1 month. Post-hoc comparisons will be performed using the Tukey test. All of the statistical analyses will be completed in the Statistical Package for Social Science (SPSS) 22 and GraphPad Prism 7.02; p < 0.05 will be considered statistically significant.